CLINICAL TRIAL: NCT00005851
Title: Phase I/II Study of HLA-Matched Non-Myeloablative Peripheral Blood Mobilized Hematopoietic Progenitor Cell Transplantation as Treatment for Patients With Metastatic Renal Cell Carcinoma. A Multi-Center Trial.
Brief Title: Low-Dose Total-Body Irradiation and Fludarabine Phosphate Followed By Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Stage IV Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1495.00; NCI-2012-00581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1495.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — fludarabine phosphate; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nonmyeloablative donor PBSC transplantation) (Experimental): CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo low-dose TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplant on day 0.
  IMMUNOSUPRESSION: Patients receive cyclosporine PO BID or IV QD or BID on days -3 to 35 with taper to day 56, and mycophenolate mofetil PO or IV over 2 hours TID on days 0-40.
  DLI: Patients with stable mixed chimerism on day 56 with no evidence of GVHD may receive escalating doses of non-mobilized DLI over 30 minutes. Patients may receive up to 4 DLIs at escalating doses if there is disease progression with no evidence of GVHD.
  Interventions: Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Procedure: peripheral blood stem cell transplantation; Biological: therapeutic allogeneic lymphocytes; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo nonmyeloablative allogeneic PBSC transplantation
Drug: cyclosporine — Given PO or IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO or IV
  Other Names: Cellcept; MMF
Procedure: peripheral blood stem cell transplantation — Undergo nonmyeloablative allogeneic PBSC transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Biological: therapeutic allogeneic lymphocytes — Undergo DLI
  Other Names: ALLOLYMPH
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The reason for doing this study is to see if cancer will respond to immune therapy after transplantation of blood stem cells (from the bone marrow) using a new kind of treatment regimen that is less toxic than that previously used for blood stem cell transplants. This type of transplant uses much less chemotherapy and radiation than standard bone marrow transplants. The treatment consists of medications that weaken the immune system so it doesn't reject the donor's marrow cells. Researchers hope that the immune cells from the donor will attack the tumor. This is called a "graft versus tumor" effect and has been seen in other types of cancer. In addition, 65 days or more after the transplant the patient may be eligible for an immune treatment that uses additional immune cells from the donor to increase the effect of the stem cells against the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether mixed or full donor hematopoietic chimerism can be safely established using a non-myeloablative conditioning regimen.

II. To determine whether mixed chimerism can be safely converted to full donor hematopoietic chimerism by infusions of donor lymphocytes (DLI).

III. To evaluate potential efficacy of this approach as a treatment for metastatic renal cancer.

OUTLINE:

CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and undergo low-dose total-body irradiation (TBI) on day 0.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplant on day 0.

IMMUNOSUPRESSION: Patients receive cyclosporine orally (PO) twice daily (BID) or IV once daily (QD) or BID on days -3 to 35 with taper to day 56, and mycophenolate mofetil PO or IV over 2 hours thrice daily (TID) on days 0-40.

DLI: Patients with stable mixed chimerism on day 56 with no evidence of graft-vs-host disease (GVHD) may receive escalating doses of non-mobilized DLI over 30 minutes. Patients may receive up to 4 DLIs at escalating doses if there is disease progression with no evidence of GVHD.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed stage IV renal cancer who have stable (including those rendered to be in remission) or progressive disease
* Human lymphocyte antigen (HLA) genotypically identical related donor willing to undergo leukapheresis initially for collection of peripheral blood stem cells (PBSC) and subsequently for collection of peripheral blood mononuclear cells (PBMC)
* Ionized calcium level within normal limits
* DONOR: HLA genotypically identical family member (excluding identical twins)
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)
* DONOR: Age < 75 years

Exclusion Criteria:

* Patients who have positive serologies for human immunodeficiency virus (HIV)1 and 2, human T-lymphotropic virus (HTLV)-1
* Patients unwilling to use contraceptive techniques during and for 12 months following treatment
* Serum creatinine > 2.0; the Fred Hutchinson Cancer Research Center (FHCRC) Patient Care Conference (PCC) may approve patients with elevated serum creatinine following presentation and approval; centers outside the FHCRC that have a PCC or equivalent should obtain their institutional approval; if there is not a comparable group at the institution, please contact the FHCRC Principal Investigator for FHCRC approval through PCC
* Cardiac ejection fraction < 50%; ejection fraction is required if the patient has a history of anthracyclines or history of cardiac disease
* Diffusion capacity of carbon monoxide (DLCO) < 50% of predicted, total lung capacity (TLC) < 50%, forced expiratory volume in one second (FEV1) < 50%
* Liver function tests including total bilirubin, serum glutamate pyruvate transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) > 2 x the upper limit of normal unless due to the malignancy
* Karnofsky score < 80
* Brain metastasis
* Ongoing active bacterial, viral or fungal infection
* Pregnancy or breastfeeding
* Patients with other active non-hematologic malignancies (except non-melanoma skin cancers)
* Patients with a history of other non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* The addition of cytotoxic agents for "cytoreduction" with the exception of Gleevec (imatinib mesylate), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or rituxan will not be allowed within three weeks of the initiation of conditioning
* DONOR: Age less than 12 years
* DONOR: Pregnancy
* DONOR: Infection with HIV
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness
* DONOR: Failure to meet criteria for donation as described in the Standard Practice Guidelines of the institution

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2000-02; Primary Completion 2004-07 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
True response rate (complete response [CR] or partial response [PR]) greater than the 15% achievable with standard therapy | Up to 5 years
  If 6 or more out of 25 patients achieve a CR or PR, then there is at least 80% confidence that the true response rate exceeds 15% and that this approach is potentially efficacious.
Transplant-related mortality | Within 200 days of transplant
  Defined as death before day 200 not related to progression of disease.
Rate of grade IV acute GVHD | Up to 90 days after last T-cell infusion

SECONDARY OUTCOMES:
Survival | Up to 5 years
  Will be examined separately and reported in a descriptive manner and confidence intervals will be presented.
Incidence of relapse | Up to 5 years
  Will be examined separately and reported in a descriptive manner and confidence intervals will be presented.
Incidence of myelosuppression after initial PBSC infusion | Up to 2 months post-transplant
  Defined as absolute neutrophil count < 500 for > 2 days, platelets < 20,000 for > 2 days. Will be examined separately and reported in a descriptive manner and confidence intervals will be presented.
Incidence of aplasia after DLI | Until 2 months post-transplant
  Will be examined separately and reported in a descriptive manner and confidence intervals will be presented.
Incidence of grades 2-4 acute GVHD after DLI | Up to 90 days after last T-cell infusion
  Will be examined separately and reported in a descriptive manner and confidence intervals will be presented.
Incidence of grades chronic extensive GVHD after DLI | Up to 90 days after last T-cell infusion
  Will be examined separately and reported in a descriptive manner and confidence intervals will be presented for all estimates.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (6):
- United States (6):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Baylor University Medical Center, Dallas, Texas
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin